CLINICAL TRIAL: NCT05953181
Title: Neoadjuvant Chemoradiotherapy Followed by Surgery Versus Active Surveillance for Oesophageal Cancer (SANO-trial): a Phase-III Stepped-wedge Cluster Randomised Trial
Brief Title: Statistical Analysis Plan for the SANO-trial: Neoadjuvant Chemoradiotherapy Followed by Surgery Versus Active Surveillance for Oesophageal Cancer
Acronym: SANO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Jan van Lanschot, prof. dr., Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC 17-392
Record Dates: First submitted 2023-07-03; First posted 2023-07-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Esophageal Cancer; Active Surveillance; Neoadjuvant Chemoradiotherapy; Surgical Oncology
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active surveillance (Experimental)
  Interventions: Procedure: Active surveillance
- Standard esophagectomy (Active Comparator)
  Interventions: Procedure: Active surveillance

INTERVENTIONS:
Procedure: Active surveillance — Patients enrolled in the active surveillance arm will undergo diagnostic evaluations every 3 months in the first year after completion of neoadjuvant treatment, every 4 months in the second year, every 6 months in the third year and yearly in the 4th and 5th year of follow up, or when symptoms or results of any diagnostic test require shorter assessment intervals. In the active surveillance arm, surgical resection will be offered only to those patients, in whom a locoregional regrowth is highly suspected or proven, without any signs of distant dissemination.

SUMMARY:
An active surveillance approach is proposed after completion of neoadjuvant chemoradiotherapy (nCRT) for carcinoma of the oesophagus. In this SANO (i.e. Surgery As Needed for Oesophageal cancer) approach, surgical resection is offered only to patients in whom a locoregional regrowth is highly suspected or proven, without distant dissemination. Such an organ-preserving strategy can have great advantages, but is only justified if long-term survival is non-inferior to that of the current standard trimodality approach comprising neoadjuvant chemoradiotherapy followed by standard surgery. The aim of this study is to assess the (cost-)effectiveness (including non-financial costs and survival) of active surveillance for patients with squamous cell- or adenocarcinoma of the oesophagus or oesophago-gastric junction.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent or are planned to undergo neoadjuvant chemoradiotherapy according to CROSS and are planned to undergo potentially curative surgical resection for histologically proven oesophageal or junctional squamous cell carcinoma or adenocarcinoma are eligible. Whenever pathology is inconclusive but a multidisciplinary expert group concludes oesophageal carcinoma because of radiologically or endosonographically highly suspected lesions, patients are eligible for the study.
* Age ≥18;
* Written, voluntary, informed consent.

Exclusion Criteria:

* Language difficulty, dementia or altered mental status prohibiting the understanding and giving of informed consent and to complete quality of life questionnaires;
* Non-FDG-avid tumour at baseline PET-CT scan;
* Initial treatment with endoscopic resection.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 776 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | the interval between the moment of achieving cCR (i.e. the moment the patient will start the intervention) and death or last follow-up, with a minimal follow-up of two years after reaching cCR.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, University Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT05953181/SAP_000.pdf